CLINICAL TRIAL: NCT01505868
Title: An Open Label Phase I/II Study of Cabazitaxel With or Without Carboplatin in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Cabazitaxel With or Without Carboplatin in Treating Patients With Previously Treated Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0727; NCI-2012-00059 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011-0727 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2011-12-30; First posted 2012-01-09 (Estimated); Results first posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Castration Levels of Testosterone; Castration-Resistant Prostate Carcinoma; Lymphadenopathy; Metastatic Prostate Carcinoma; Prostate Adenocarcinoma; Prostate Carcinoma Metastatic in the Bone; Prostate Small Cell Carcinoma
MeSH Terms: conditions — Lymphadenopathy; Prostatic Neoplasms | interventions — cabazitaxel; XRP6258; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (cabazitaxel) (Experimental): Patients receive cabazitaxel IV over 60-90 minutes on day 1. Treatment repeats every 21 days for up to 10 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabazitaxel; Other: Laboratory Biomarker Analysis
- Arm II (cabazitaxel and carboplatin) (Experimental): Patients receive cabazitaxel IV over 60-90 minutes and carboplatin IV over 60-90 minutes on day 1. Treatment repeats every 21 days for up to 10 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabazitaxel; Drug: Carboplatin; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cabazitaxel — Given IV
  Other Names: Jevtana; RPR-116258A; Taxoid XRP6258; XRP-6258
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm II (cabazitaxel and carboplatin)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This partially randomized phase I/II trial studies cabazitaxel with or without carboplatin in treating patients with previously treated prostate cancer that has spread to other areas of the body and does not respond to treatment with hormones. Drugs used in chemotherapy, such as cabazitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving cabazitaxel alone or with carboplatin is more effective in treating prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dosage (MTD) of cabazitaxel-carboplatin in the phase I portion of the study.

II. To evaluate progression free survival achieved with cabazitaxel-carboplatin versus cabazitaxel alone in men with metastatic castration resistant prostate cancer (mCRPC) in the phase II portion of the study.

SECONDARY OBJECTIVES:

I. To assess prostate-specific antigen (PSA) response rate (percentage of patients with > 50 % decline).

II. To correlate changes in bone specific alkaline phosphatase and urine n-telopeptides with response.

III. To evaluate overall survival. IV. To evaluate safety and toxicity. V. To evaluate influence of the anaplastic phenotype on response to therapy. VI. To collect and archive serum, plasma, and urine samples in study patients for later hypothesis generating associations.

OUTLINE: This is a phase I, dose-escalation study followed by a randomized phase II study.

PHASE I: Patients receive cabazitaxel intravenously (IV) over 60-90 minutes and carboplatin IV over 60-90 minutes on day 1. Treatment repeats every 21 days for up to 10 courses in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cabazitaxel IV over 60-90 minutes on day 1. Treatment repeats every 21 days for up to 10 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive cabazitaxel IV over 60-90 minutes and carboplatin IV over 60-90 minutes on day 1. Treatment repeats every 21 days for up to 10 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic evidence of prostate adenocarcinoma
* In addition to patients with adenocarcinoma, patients with "anaplastic" features are also eligible as defined by at least one of the following: a) histologic evidence of small cell prostate cancer (patients with small cell carcinoma on histology are not required to demonstrate castration-resistant progression); b) any of the following metastatic presentations: (i) exclusive visceral metastases; (ii) radiographically predominant lytic bone metastases identified by plain X-ray or computed tomography (CT) scan; (iii) bulky (>= 5 cm in longest dimension) lymphadenopathy (iv) bulky (>= 5 cm) tumor mass in the prostate/pelvis (v) low PSA (=< 10 ng/ml) at initial presentation (prior to androgen ablation or at symptomatic progression in the castrate-setting) plus high volume (>= 20) bone metastases; (vi) elevated serum lactate dehydrogenase (LDH) (>= 2 x ULN) or elevated serum carcinoembryonic antigen (CEA) (>= 2 x upper limit of normal [ULN]) in the absence of other etiologies; (vii) short interval (=< 180 days) to castrate-resistant progression following initiation of hormonal therapy
* Castration-resistant prostate cancer; patients must have surgical or ongoing chemical castration (with luteinizing-hormone-releasing hormone [LHRH] agonists or LHRH antagonists), with a baseline testosterone level < 50 ng/dL
* Metastatic disease; patients must have evidence for metastatic prostate cancer by bone scan and/or CT/magnetic resonance imaging (MRI) (i.e., soft tissue, visceral, lymph node); if lymph node, visceral and/or soft-tissue metastases are the only evidence of metastasis, at least one lesion must be >= 1.5 cm in diameter
* Patients may have received prior treatment with androgen ablative therapies (such as bicalutamide, ketoconazole, diethylstilbestrol [DES], abiraterone, Xtandi, ARN-509) and/or "targeted" therapies (such as tyrosine kinase inhibitors); androgen ablative therapies must be discontinued >= 3 days prior to initiation of study treatment with the exception of abiraterone and/or enzalutamide, which may be continued during study treatment per the practice preference of the treating physician; patients who are predicted to benefit from an antiandrogen withdrawal response should be tested for this possibility before being considered for eligibility to this study; targeted therapies must be discontinued >= 2 weeks before initiation of study treatment
* Both chemotherapy-naive and patients previously treated with chemotherapy are eligible; chemotherapy pretreated patients may have received a maximum of two prior systemic cytotoxic chemotherapies completed at least 3 weeks prior to initiation of study treatment
* Patients must have documented evidence of progressive disease as defined by any of the following: a) PSA progression: minimum of 2 rising values (3 measurements) obtained a minimum of 7 days apart with the last result being at least >= 2.0 ng/mL; b) new or increasing non-bone disease (by Response Evaluation Criteria In Solid Tumors [RECIST]); c) positive bone scan with 2 or more new lesions (Prostate Cancer Working Group [PCWG2])
* For purposes of stratification, patients will be categorized as "responders" or "non-responders" based on their response to prior docetaxel-based therapy; a) responders will have demonstrated objective responses to first-line docetaxel as determined by any of the following: 1. decrease in PSA level >= 50% from baseline, maintained for >= 6 weeks; 2. partial or complete response in lymph nodes and soft tissue metastases by RECIST; responders must have received >= 225 mg/m^2 (~ 3 cycles) of docetaxel; b) patients not meeting response criteria above will be considered as non-responders; we anticipate 2 general categories of non-responders based on the following disease phenotypes: 1. progressive disease on therapy without any objective evidence of response ("primary-resistant disease"); progressive disease on therapy with prior objective evidence of response, but response duration is =< 6 weeks ("docetaxel refractory disease"); non-responders are eligible even if they have received < 225 mg/m^2 of docetaxel
* If present, peripheral neuropathy must be =< grade 2
* Absolute neutrophil count (ANC) >= 1,500/ml (unless due to bone marrow infiltration by tumor in which case ANC >= 500/ml are allowed) (within 14 days before registration)
* Platelets >= 100,000/ml (unless due to bone marrow infiltration by tumor in which case >= 50,000/ml are allowed) (within 14 days before registration)
* Total bilirubin =< upper limit of normal with the exception of isolated hyperbilirubinemia due to Gilbert's syndrome or if the patient has liver metastases and/or acute tumor-associated illness =< 4 x ULN (within 14 days before registration)
* Serum glutamic-pyruvic transaminase (SGPT), (alanine aminotransferase [ALT]) AND/OR serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 1.5 x the ULN or if patient has liver metastases and/or acute tumor-associated illness, =< 4 x ULN (within 14 days before registration)
* Patient has creatinine clearance >= 30 ml/min using the Cockcroft-Gault equation (within 14 days before registration)
* Men whose partner is a woman of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter
* Patient or his legally authorized representative must provide written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2

Exclusion Criteria:

* Radiation therapy (including palliative radiotherapy to a metastatic lesion) within 14 days or major surgery (e.g., open abdominal, pelvic, thoracic, orthopedic or neurosurgery) within 28 days of the date of the first dose
* Samarium-153 within 28 days of registration, or strontium-89 within 12 weeks (84 days) of registration; patients who have received 2 or more doses of bone-seeking radioisotopes are not eligible
* Current treatment on another therapeutic clinical trial
* Prior treatment with cabazitaxel and/or carboplatin
* Impending complication from bone metastases (fracture and/or cord compression); properly treated or stabilized fractures and/or cord compression is allowed
* Presence of ongoing urinary obstruction (e.g., urinary retention, hydronephrosis) requiring medical intervention; properly treated urinary obstruction is allowed
* Patient has an uncontrolled intercurrent illness (e.g., uncontrolled diabetes, uncontrolled hypertension)
* Patient has another serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the patient's ability to provide informed consent or with the completion of treatment according to this protocol
* Patients with a history of severe hypersensitivity reaction to JEVTANA® (cabazitaxel) or other drugs formulated with polysorbate 80
* Patients with an active second malignancy that could, in the investigator's opinion, potentially interfere with the patient's ability to participate and/or complete this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-07-11 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Corn, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Corn PG, Heath EI, Zurita A, Ramesh N, Xiao L, Sei E, Li-Ning-Tapia E, Tu SM, Subudhi SK, Wang J, Wang X, Efstathiou E, Thompson TC, Troncoso P, Navin N, Logothetis CJ, Aparicio AM. Cabazitaxel plus carboplatin for the treatment of men with metastatic castration-resistant prostate cancers: a randomised, open-label, phase 1-2 trial. Lancet Oncol. 2019 Oct;20(10):1432-1443. doi: 10.1016/S1470-2045(19)30408-5. Epub 2019 Sep 9. PMID 31515154
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were treated at MD Anderson Cancer Center in Houston, TX and Karmanos Cancer institute in Detroit, MI
Pre-assignment Details: 170 participants enrolled, 10 were phase I participants, 1 participant withdrew in phase I
Groups:
- Phase I Cabazitaxel + Carboplatin Dose Zero: Intravenous cabazitaxel 20 mg/m2 and carboplatin area under the curve (AUC) 3 mg/mL per min every 21 days
- Phase I Cabazitaxel + Carboplatin Dose One: Intravenous cabazitaxel 20 mg/m2 and carboplatin area under the curve (AUC) 4 mg/mL per min every 21 days
- Phase I Cabazitaxel + Carboplatin Dose Two: Intravenous cabazitaxel 25 mg/m2 and carboplatin area under the curve (AUC) 4 mg/mL per min every 21 days
- Phase II Cabazitaxel: Intravenous cabazitaxel 25 mg/m2 every 21 days up to 10 doses
- Phase II Cabazitaxel + Carboplatin: Intravenous cabazitaxel 25 mg/m2 and carboplatin AUC 4 every 21 days up to 10 doses
Period: Overall Study
Arm/Group | Phase I Cabazitaxel + Carboplatin Dose Zero | Phase I Cabazitaxel + Carboplatin Dose One | Phase I Cabazitaxel + Carboplatin Dose Two | Phase II Cabazitaxel | Phase II Cabazitaxel + Carboplatin
Started | 4 | 3 | 3 | 79 | 81
Completed | 3 | 3 | 3 | 79 | 81
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I Cabazitaxel + Carboplatin Dose Zero: Intravenous cabazitaxel 20 mg/m2 and carboplatin AUC 3 every 21 days up to 10 doses
- Phase I Cabazitaxel + Carboplatin Dose One: Intravenous cabazitaxel 20 mg/m2 and carboplatin AUC 4 every 21 days up to 10 doses
- Phase I Cabazitaxel + Carboplatin Dose Two; Phase II Cabazitaxel + Carboplatin: Intravenous cabazitaxel 25 mg/m2 and carboplatin AUC 4 every 21 days up to 10 doses
- Total: Total of all reporting groups
Arm/Group | Phase I Cabazitaxel + Carboplatin Dose Zero | Phase I Cabazitaxel + Carboplatin Dose One | Phase I Cabazitaxel + Carboplatin Dose Two | Phase II Cabazitaxel | Phase II Cabazitaxel + Carboplatin | Total
Number analyzed (Participants) | 3 | 3 | 3 | 79 | 81 | 169
Age, Continuous [Mean (Full Range); unit: years] | 66 [55 to 77] | 74 [72 to 78] | 69 [66 to 72] | 66 [61 to 69] | 68 [62 to 73] | 67 [61 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 79 | 81 | 169
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 4 | 8 | 13
  Not Hispanic or Latino | 0 | 0 | 0 | 12 | 18 | 30
  Unknown or Not Reported | 2 | 3 | 3 | 63 | 55 | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 16 | 8 | 24
  White | 3 | 3 | 3 | 57 | 64 | 130
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 6 | 9 | 15
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 79 | 81 | 169
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — Grade 0: Fully active, able to carry on all pre-disease performance without restriction. Grade 1: Restricted in physically strenuous activity but ambulatory, able to carry out light house work, office work. Grade 2: Ambulatory and capable of all selfcare but unable to carry out any work activities awake at least 50% of day.
  Participants
    Grade 0 | 1 | 1 | 1 | 21 | 22 | 46
    Grade 1 and 2 | 2 | 2 | 2 | 58 | 59 | 123
Prostate-specific antigen (PSA) [Mean (Full Range); unit: µg/L] | 380.4 [21.1 to 653.3] | 89.5 [27 to 160] | 217.6 [6.7 to 551.8] | 23.7 [8.6 to 81.2] | 33.8 [11.4 to 146.3] | 28.75 [8.6 to 146.3]
Bone metastases [Count of Participants; unit: Participants]
  No | 0 | 0 | 0 | 7 | 6 | 13
  Yes | 3 | 3 | 3 | 72 | 75 | 156

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dosage (MTD) of Cabazitaxel-carboplatin in the Phase I Portion of Study
Description: The MTD was defined as the highest dose cohort studied in which one of six or fewer patients experienced a dose-limiting toxicity.
Time Frame: 6 months
Measure: Number; unit: mg/m^2
Groups:
- Phase I Cabazitaxel + Carboplatin: Intravenous cabazitaxel 25 mg/m2 and carboplatin area under the curve (AUC) 4 mg/mL per min every 21 days
Arm/Group | Phase I Cabazitaxel + Carboplatin
Number analyzed (Participants) | 9
mg/m^2 | 25

2. Primary Outcome: Progression Free Survival (PFS) of Cabazitaxel-carboplatin Versus Cabazitaxel in the Phase II Portion of Study
Description: PFS is the time from the first dose until progression of disease or death, whichever comes first. PFS times will be estimated using the Kaplan-Meier method.
Time Frame: From the first dose until progression of disease or death, whichever comes first, up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II Cabazitaxel | Phase II Cabazitaxel + Carboplatin
Number analyzed (Participants) | 79 | 81
months | 4.5 [3.5 to 5.7] | 7.3 [5.5 to 8.2]

3. Secondary Outcome: Prostate Specific Antigen (PSA) Response Rate
Description: Percentage of participants with a greater than 50% decrease in measurable values of PSA during treatment from their baseline PSA.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II Cabazitaxel | Phase II Cabazitaxel + Carboplatin
Number analyzed (Participants) | 66 | 68
percentage of participants | 40.9 [30.2 to 51.8] | 61.7 [51.4 to 72.6]

4. Secondary Outcome: Bone-Specific Alkaline Phosphatase Response
Description: Percentage of participants with a greater than 50% decrease in measurable values of bone-specific alkaline phosphatase during treatment from their baseline values
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II Cabazitaxel | Phase II Cabazitaxel + Carboplatin
Number analyzed (Participants) | 34 | 50
percentage of participants | 29.4 [19 to 39] | 62 [51.4 to 72.6]

5. Secondary Outcome: Urine N-Telopeptides Response
Description: Percentage of participants with a greater than 50% decrease in measurable values of urine n-telopeptides during treatment from their baseline values.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II Cabazitaxel | Phase II Cabazitaxel + Carboplatin
Number analyzed (Participants) | 20 | 24
percentage of participants | 55 [33.2 to 76.8] | 62.5 [42.1 to 81.9]

6. Secondary Outcome: Overall Survival (OS)
Description: Time from date of treatment start until date of death due to any cause or last follow up.
Time Frame: Time from date of treatment start until date of death due to any cause or last follow up, up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II Cabazitaxel | Phase II Cabazitaxel + Carboplatin
Number analyzed (Participants) | 79 | 81
months | 17.3 [13.8 to 21.9] | 18.5 [16.7 to 21.9]

7. Secondary Outcome: Phase II Most Common Grade 3-5 Adverse Events
Description: Grade 3: Serious reaction which requires medical treatment Grade 4: Life threatening. Grade 5 Death.
Time Frame: Time from date of treatment start until date of death due to any cause or last follow up, up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Cabazitaxel | Phase II Cabazitaxel + Carboplatin
Number analyzed (Participants) | 79 | 81
Participants
  Fatique | 9 | 20
  Anemia | 4 | 23
  Neutropenia | 4 | 16
  Thrombocytopenia | 1 | 14

8. Post Hoc Outcome: Aggressive Variant Prostate Carcinoma-Metastatic (ACPC-MS) Phenotypes Correlated to Response
Description: PFS and OS were reported for participants with and without AVPC-MS in the cabazitaxel vs cabazitaxel + carboplatin treatment groups
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- AVPC-MS Postive: Immunochemistry positive for AVPC-MS
- AVPC-MS Negative: Immunochemistry negative for AVPC-MS
Arm/Group | AVPC-MS Postive | AVPC-MS Negative
Number analyzed (Participants) | 26 | 30
months
  Cabazitaxel PFS | 1.7 [1.3 to NA] — below the level of detection | 6.3 [5.9 to 10.9]
  Cabazitaxel + carboplatin PFS | 7.5 [4.4 to 9.6] | 6.5 [3.9 to 8.4]
  Cabazitaxel OS | 8.5 [4.8 to NA] — below the level of detection | 21.7 [17.4 to NA] — below the level of detection
  Cabazitaxel + carboplatin OS | 20.2 [13.3 to 37.2] | 21.5 [9.1 to NA] — below the level of detection

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- Phase I Cabazitaxel + Carboplatin Dose Zero: Intravenous cabazitaxel 20mg/m2 and carboplatin area under the curve (AUC) 3mg/mL per min every 21 days
Arm/Group | Phase I Cabazitaxel + Carboplatin Dose Zero | Phase I Cabazitaxel + Carboplatin Dose One | Phase I Cabazitaxel + Carboplatin Dose Two | Phase II Cabazitaxel | Phase II Cabazitaxel + Carboplatin
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 63/79 | 69/81
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 3/79 | 4/81
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 78/79 | 81/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Cabazitaxel + Carboplatin Dose Zero (N=3) | Phase I Cabazitaxel + Carboplatin Dose One (N=3) | Phase I Cabazitaxel + Carboplatin Dose Two (N=3) | Phase II Cabazitaxel (N=79) | Phase II Cabazitaxel + Carboplatin (N=81)
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 1 (1)
Fever (General disorders) | 0 | 0 | 0 | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (2) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 | 0 | 0 | 0 (0) | 1 (1)
WBC decreased (Investigations) | 0 | 0 | 0 | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Cabazitaxel + Carboplatin Dose Zero (N=3) | Phase I Cabazitaxel + Carboplatin Dose One (N=3) | Phase I Cabazitaxel + Carboplatin Dose Two (N=3) | Phase II Cabazitaxel (N=79) | Phase II Cabazitaxel + Carboplatin (N=81)
Gastrointestinal disorders (Gastrointestinal disorders) | 0 | 0 | 0 | 4 (7) | 7 (8)
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 4 (4) | 4 (4)
Alkaline phosphatase increased (Investigations) | 2 | 0 | 0 | 3 (3) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 14 (14) | 24 (26)
Anemia (Blood and lymphatic system disorders) | 2 | 1 | 3 | 20 (31) | 47 (112)
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 7 (7) | 17 (21)
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 2 (2) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 5 (5) | 12 (14)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 (2) | 7 (8)
Bruising (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 (1) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 14 (23) | 35 (58)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 (3) | 4 (6)
Creatinine increased (Investigations) | 0 | 1 | 2 | 7 (8) | 8 (11)
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1 | 2 (2) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 4 (4) | 8 (12)
Diarrhea (Gastrointestinal disorders) | 0 | 3 | 2 | 44 (102) | 54 (160)
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 6 (6) | 13 (16)
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 11 (11) | 16 (22)
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 19 (34) | 34 (71)
Edema limbs (General disorders) | 1 | 1 | 1 | 11 (13) | 10 (13)
Epitaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (2) | 6 (8)
Fatigue (General disorders) | 1 | 3 | 3 | 58 (125) | 69 (272)
Fever (General disorders) | 1 | 1 | 0 | 5 (5) | 9 (14)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 (10) | 3 (3)
Flu like symptoms (General disorders) | 0 | 0 | 0 | 1 (1) | 6 (8)
Flushing (Vascular disorders) | 0 | 0 | 0 | 3 (5) | 4 (4)
Genralized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (2) | 5 (7)
Headache (Nervous system disorders) | 0 | 0 | 1 | 6 (10) | 7 (7)
Hematuria (Renal and urinary disorders) | 1 | 0 | 0 | 3 (4) | 10 (14)
Hemoglobinuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 (1) | 5 (5)
Hot flashes (Vascular disorders) | 0 | 0 | 1 | 3 (3) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 (1) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 14 (17) | 16 (24)
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 3 (3) | 6 (11)
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 6 (7) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 3 (3) | 5 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 5 (6) | 10 (18)
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 7 (9) | 13 (31)
Hypomagnesenia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 6 (7) | 35 (51)
Hyponatrenia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 (5) | 6 (7)
Hypotension (Vascular disorders) | 1 | 0 | 0 | 2 (3) | 6 (9)
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 5 (6) | 2 (2)
Localized Edema (General disorders) | 1 | 0 | 0 | 1 (1) | 3 (3)
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 9 (17) | 8 (19)
Malaise (General disorders) | 0 | 0 | 0 | 1 (1) | 8 (9)
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 6 (11) | 7 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 (4) | 4 (6)
Nausea (Gastrointestinal disorders) | 0 | 2 | 2 | 28 (60) | 57 (170)
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 6 (7) | 16 (32)
Non-cardiac cest pain (General disorders) | 1 | 0 | 1 | 4 (5) | 1 (1)
Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 7 (14) | 9 (9)
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3 (4) | 8 (11)
Paresthesia (Nervous system disorders) | 0 | 1 | 0 | 8 (10) | 15 (18)
Neuropathy (Nervous system disorders) | 0 | 1 | 1 | 5 (8) | 16 (23)
Platelet count decreased (Investigations) | 2 | 1 | 0 | 5 (7) | 32 (83)
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 1 (1) | 6 (7)
Urinary urgency (Renal and urinary disorders) | 0 | 1 | 0 | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 4 (4) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 14 (25) | 30 (63)
Weight loss (Investigations) | 1 | 0 | 0 | 4 (5) | 12 (14)
WBC decreased (Investigations) | 0 | 0 | 0 | 8 (11) | 24 (50)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT01505868/Prot_SAP_000.pdf